CLINICAL TRIAL: NCT01781065
Title: The Analgesic Effect of Transcranial Direct Current Stimulation Over the Primary Motor Cortex on Central Neuropathic Pain Patients With Spinal Cord Injury
Brief Title: The Effects of Transcranial Direct Current Stimulation on Central Pain in Patients With Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Ik Shin, Associate Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-2008-010 SNUBH
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Neuropathic Pain; Spinal Cord Injury
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- transcranial direct current stimulation (Experimental): Anodal stimulation on motor cortex
  Interventions: Device: transcranial direct current stimulation
- Sham transcranial direct current stimulation (Sham Comparator): Turn off after 10 s of stimulation
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation
  Other Names: Iomed Phoresor II Auto

SUMMARY:
The purpose of this study is to evaluate the analgesic effect of transcranial direct current stimulation (tDCS) applied on motor cortex in patients with spinal cord injury who have chronic neuropathic pain.

DETAILED DESCRIPTION:
* anodal stimulation of the primary motor cortex (M1)
* anode electrode: C3 (EEG 10/20 system)
* cathode electrode: contralateral supraorbital area
* constant current of 2mA intensity for 20 min
* twice a day with a more than 4 hours interval during of 2 weeks (from Monday to Friday, total 20 treatment session)

ELIGIBILITY:
Inclusion Criteria:

* elapsed time since spinal cord injury more than 6 months
* stable chronic pain for at least 3 preceding months
* pain that was not attributable to cause other that neuropathic pain
* pain that was resistant to various types of medications or physical or complementary medicine treatment

Exclusion Criteria:

* any kind of metal implant in the head
* heart disease including having a cardiac maker
* family or personal history of epilepsy, or neuropsychiatric illness

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale for average pain over the preceding 24h | before the first tDCS session, and 1, 2, 4, 6 and 8 wk after the start of the stimulation

SECONDARY OUTCOMES:
Patient global impression of change for pain | before the first tDCS session, and 1, 2, 4, 6, and 8 wk after the start of the stimulation

OTHER OUTCOMES:
Pain interference in general daily life, mood and sleep | before the first tDCS session, and 1, 2, 4, 6, 8 wk after start of the stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Ik Shin, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618